CLINICAL TRIAL: NCT05643430
Title: A Prospective Multicenter Single Arm Trial to Assess the Safety and Effectiveness of Additional Sizes of the BioFreedom Ultra CoCr Biolimus A9 Coated Coronary Stent System
Brief Title: ULTRA LONG: BioFreedom Ultra
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biosensors Europe SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-EU-02
Record Dates: First submitted 2022-10-28; First posted 2022-12-08 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Coronary Artery Disease; High Bleeding Risk Patients
Keywords: BioFreedom Ultra
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, open-label single-arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BioFreedom Ultra (Experimental): All patients will receive the BioFreedom Ultra as per treatment.
  Interventions: Device: BioFreedom Ultra

INTERVENTIONS:
Device: BioFreedom Ultra — The BioFreedom Ultra CoCr DCS is a combination product consisting of two key components: the cobalt chromium stent platform coated abluminally with the active ingredient BA9TM (polymer and carrier free) and the delivery system.

SUMMARY:
The goal of this Prospective, multi-center, open-label single-arm study is to Assess the Safety and Effectiveness of additional sizes of the BioFreedom Ultra CoCr Biolimus A9 coated coronary stent system in Patients at high risk of bleeding (HBR). The main question it aims to answer is to evaluate if the additional sizes of the BioFreedom Ultra have corresponding clinical safety and efficacy characteristics as the regulatory approved (=CE Marked) sizes.

ELIGIBILITY:
Clinical:

1. Patients at high bleeding risk (HBR) with an indication for PCI. This includes subjects with chronic coronary syndrome, unstable angina, or non-ST elevation myocardial infarction.
2. Patients must provide written informed consent
3. Patient is at least 18 years old
4. Patients with a life expectancy of > 1 year at time of consent
5. HBR patients defined according to the ARC-HBR criteria and suitable to receive dual anti platelet therapy (DAPT) for one month. To be qualified HBR, patients have to have at least 1 major and/or 2 minor criteria defined as follow:

   Major Minor Age ≥75 years old Anticipated use of long-term oral anticoagulation* Severe or end-stage CKD (eGFR <30 mL/min) Moderate CKD (eGFR 30-59 mL/min) Hemoglobin <11 g/dL Hemoglobin 11-12.9 g/dL for men and 11-11.9 g/dL for women Spontaneous bleeding requiring hospitalization or transfusion in the past 6 months or at any time, if recurrent Spontaneous bleeding requiring hospitalization or transfusion within the past 12 months not meeting the major criterion Moderate or severe baseline thrombocytopenia† (platelet count <100×109/L) Chronic bleeding diathesis Liver cirrhosis with portal hypertension Long-term use of oral NSAIDs or steroids Active malignancy‡ (excluding non-melanoma skin cancer) within the past 12 months Previous spontaneous ICH (at any time) Previous traumatic ICH within the past 12 months Presence of a bAVM Moderate or severe ischemic stroke§ within the past 6 months Any ischemic stroke at any time not meeting the major criterion Nondeferrable major surgery on DAPT Recent major surgery or major trauma within 30 days before PCI bAVM indicates brain arteriovenous malformation; CKD, chronic kidney disease; DAPT, dual antiplatelet therapy; eGFR, estimated glomerular filtration rate; HBR, high bleeding risk; ICH, intracranial hemorrhage; NSAID, nonsteroidal anti-inflammatory drug; and PCI, percutaneous coronary intervention.

   *This excludes vascular protection doses.

   †Baseline thrombocytopenia is defined as thrombocytopenia before PCI.

   ‡Active malignancy is defined as diagnosis within 12 months and/or ongoing requirement for treatment (including surgery, chemotherapy, or radiotherapy).

   §National Institutes of Health Stroke Scale score ≥5.

   Angiographic:
6. Patients scheduled to undergo PCI of a de novo lesion (no in-stent restenosis) with reference vessel diameter and lesion length suitable for treatment with at least one study device

Exclusion Criteria:

1. Pregnant and breastfeeding women
2. Patients lacking capacity (i.e. patients suffering from dementia and others) to provide informed consent
3. Patients not expected to comply with 1 month of DAPT
4. Staged procedures in the target vessel
5. Active bleeding at the time of inclusion
6. Cardiogenic shock
7. Unlikely compliance with long-term single anti-platelet therapy
8. Known hypersensitivity or contraindication to aspirin, clopidogrel (or to any other P2Y12 inhibitor if applicable), cobalt chromium, zinc, Biolimus A9 or a sensitivity to contrast media, which cannot be adequately pre-medicated
9. Currently participating in another trial before reaching primary endpoint
10. Patients under judicial protection, tutorship or curatorship (France only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2026-03-08 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
TLF | at 9 months after index procedure
  Incidence of Target Lesion Failure, clinically-driven target lesion revascularization (cd-TLR), Cardiovascular Death and TV-MI

SECONDARY OUTCOMES:
CD-TLR | Clinical endpoints measured at 9 and 24 months
  Incidence of Clinically driven Target Lesion Revascularization
Cardiovascular Death | Clinical endpoints measured at 9 and 24 months
  Incidence
TV-MI | Clinical endpoints measured at 9 and 24 months
  Target-Vessel Myocardial Infarction
TVR | Clinical endpoints measured at 9 and 24 months
  Target Vessel Revascularization
Stent thrombosis rate - definite/probable | Clinical endpoints measured at 9 and 24 months
  Incidence
All cause mortality | Clinical endpoints measured at 9 and 24 months
  Incidence
Bleeding rate (BARC 2-5) | Clinical endpoints measured at 9 and 24 months
  Incidence of BARC 2-5
Peri-procedural endpoints | Peri-procedural endpoints measured at 9 and 24 months
  Incidence of Device success; Lesion success and Procedure success

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Garot, Professor, Principal Investigator — Cardiovascular Institute Paris Sud (ICPS)
Locations (9):
- France (3):
  - Cardiovascular Institute Paris Sud (ICPS) L'Hôpital Privé Jacques Cartier, Massy, Massy
  - Arnault Institute Tzanck, Saint-Laurent-du-Var, Saint-Laurent-du-Var
  - Pôle Santé République, Clermont-Ferrand
- United Kingdom (6):
  - University Hospitals Birmingham (UHB), Birmingham
  - Royal Blackburn Hospital, Blackburn
  - Hull University Teaching Hospitals (HUTH), Hull
  - United Lincolnshire Hospitals (ULH), Lincoln
  - The Grange University Hospital, Newport, Newport
  - Royal Albert Edward Infirmary, Wigan

IPD SHARING:
Plan to Share IPD: Undecided